CLINICAL TRIAL: NCT06839261
Title: Efficacy and Reliability of Photo-Based Artificial Intelligence Algorithms in Assessing Difficulty of Intubation With a Double-Lumen Tube
Brief Title: Evaluation of Double Lumen Tube Intubation Difficulty With Photo-Based Artificial Intelligence Algorithms
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Onur Kucuk, Principal Investigator, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-KAEK-24/07
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Intubation; Difficult; Artificial Intelligence (AI); Double Lumen Tube Intubation
Keywords: airway management; Double lumen tube; Difficult intubation; artificial intelligence; thoracic surgery
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intubation - Difficult: According to the Intubation Difficulty Scale (IDS), a score of > 5 was defined as difficult intubation.
  Interventions: Diagnostic Test: Intubation Difficulty Scale; Other: Artificial Intelligence
- Intubation - Easy: According to the Intubation Difficulty Scale (IDS), a score of ≤ 5 was defined as easy intubation.
  Interventions: Diagnostic Test: Intubation Difficulty Scale; Other: Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Intubation Difficulty Scale — The Intubation Difficulty Scale (IDS) is an objective way to classify easy and difficult intubation. A score ≤ 5 indicates an easy or mildly difficult intubation, while IDS > 5 suggests difficult intubation, requiring additional techniques or attempts.
Other: Artificial Intelligence — The program made with Python 3 programming language using open source libraries. It will be developed to predict difficult intubation with 6 different photo data of patients, this process will be taught with a learning process and then tested.

SUMMARY:
The complexity and difficulty of intubation with double lumen tubes requires the use of advanced technologies in the management of this procedure. The potential of photo-based artificial intelligence algorithms to predict and minimize the difficulties encountered during intubation is the main motivation for this study.

The utilization of artificial intelligence algorithms within the domain of airway management holds considerable promise in providing real-time feedback to anesthesiologists, enhancing the efficacy of intubation procedures, and reducing the occurrence of complications. Specifically, photo-based AI systems can facilitate a more comprehensive understanding of airway anatomy by analyzing images captured prior to and during intubation, thereby enhancing the management of complex cases.The objective of this study is to examine the efficacy and reliability of photo-based artificial intelligence algorithms in evaluating the complexity of intubation with a double lumen tube.The integration of artificial intelligence into the intubation process is intended to enhance patient outcomes and establish a new benchmark for anesthesia practice. This study aims to address the existing gap in the literature and provide innovative approaches to clinical practice.

Informed consent was obtained from patients undergoing thoracic surgery operations, and demographic data (age, height, body weight, body mass index, gender), American Society of Anesthesiologists (ASA) score, type of operation, and comorbid diseases (diabetes mellitus, hypertension, coronary artery disease, chronic kidney disease, chronic obstructive pulmonary disease, asthma, obstructive sleep apnea) were obtained. Thoracic and/or extrath oracic malignancy history), parameters considered as risk factors for difficult intubation (history of previous difficult intubation, LEMON criteria (look externally, evaluate, mallampathy, obstruction, neck mobility), upper lip bite test) and photographs of the patients (including head and neck region) will be recorded in six different directions and ways with a professional camera (actively used in our hospital) in the preoperative period. During the intraoperative phase, the Cormack-Lehane scoring system will be employed, and the intubation process with a double-lumen tube will be evaluated for ease or difficulty. Intraoperative complications related to the operation will also be documented.The data will then be processed using Python 3 programming language and open-source libraries to calculate artificial intelligence algorithms. In the event of incomplete patient data, data imputation techniques will be employed to supplement the artificial intelligence program.

The primary outcome variable of the study is the rate at which the photo-based artificial intelligence algorithm predicts whether intubation with a double lumen tube is easy or difficult.The secondary outcome variable is the comparison of the rate of prediction of intubation with double lumen tube by photo-based artificial intelligence algorithms and the rate of prediction of intubation with double lumen tube by conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing thoracic surgery
* Giving informed consent
* Over 18 years of age
* Double lumen tube used for intubation
* ASA (American Society of Anesthesiologist)1-2-3

Exclusion Criteria:

* Emergency surgeries
* ASA 4 and above
* Head and neck tumor, history of surgery/RT related to tumor
* Presence of syndrome that will cause difficult intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was calculated as 214 patients with a power of 0.90, 5% type-1 error, 81.8% sensitivity and 26.7% prevalence (AUC=0.864) with a power of 0.90, 5% type-1 error, 81.8% sensitivity and (AUC=0.864) 26.7% prevalence in the Sample Size Estimation for Diagnostic Accuracy Studies calculated for the study considering the literature data. Since 214 patients would be used to teach the AI easy and difficult intubation and 46 patients would be used to test the AI, a total of 260 patients were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Intubation Difficulty Scale (IDS) | During the operation
  The Intubation Difficulty Scale (IDS) is an objective way to classify easy and difficult intubation. A score ≤ 5 indicates an easy or mildly difficult intubation, while IDS > 5 suggests difficult intubation, requiring additional techniques or attempts.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Küçük, Specialist, Principal Investigator — Ankara Atatürk Sanatoryum Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatoryum Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No